CLINICAL TRIAL: NCT04974593
Title: Predictive Value of Hydrogen/Methane Lactose Breath Testing on the Therapeutic Effect of Lactose-free Diet in Moderate to Severe ROME IV IBS.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: PreVaIL
Record Dates: First submitted 2021-07-13; First posted 2021-07-23 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Irritable Bowel Syndrome; Lactose Intolerant
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Results from H2 and CH4 excretion, as well as symptom scores during the breath test will remain unknown to the participants and the study personnel until the end of the study to guarantee study blinding. However, because of the imbalance in the proportion of lactose H2BT-positive vs. -negative subjects, results of the H2BT will be analyzed by a trained physician with no contact with study subjects or investigators in order to guarantee that sufficient subjects are recruited in both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- H2BT-positive (Experimental)
  Interventions: Other: low fat diet
- H2BT-negative (Experimental)
  Interventions: Other: low fat diet

INTERVENTIONS:
Other: low fat diet — A trained dietitian will provide instruction of the LFD according to standard practice.

SUMMARY:
Lactose intolerance (LI) results from lactose malabsorption (LM) secondary to insufficient hydrolysis of the disaccharide lactose into galactose and glucose (Misselwitz 2019). The undigested lactose will eventually reach the colon, resulting in fermentation from colonic bacteria with production of different compounds such as short chain fatty acids, carbon dioxide, H2 and methane (Catanzaro 2021). These compounds have an osmotic effect and can stimulate colonic contractions. These pathophysiological mechanisms encountered in patients suffering from LI generate symptoms, such as abdominal pain and cramps, flatulence, diarrhea, borborygmi among others. As dairy products are highly present in our Western diet, LI will often be considered in patients presenting with these symptoms and they will be referred for further testing. When LM is diagnosed, a lactose-free diet (LFD) will be advocated to alleviate symptoms. However, studies indicate that individuals with LM should tolerate up to 12 g of lactose when administered in a single dose (Suchy 2010).

Irritable bowel syndrome (IBS) is another frequently encountered disorder. According to the Rome IV criteria, it is characterized by abdominal pain associated with a change in stool frequency or consistency, or with symptomatic improvement by defecation (Mearin 2016). Associated symptoms, such as bloating and flatulence, are frequently reported. As such, discerning between IBS and LI based on symptoms alone can be challenging. Moreover lactose is considered part of the so-called fermentable oligo-, di-, monosaccharides and polyols (FODMAPs). A low FODMAP diet has been advocated for IBS with beneficial response in at least part of the patients (Halmos 2014).

Many studies investigated the role of lactose in IBS. These studies were performed in the pre-Rome IV era and before standardized interpretation rules for Hydrogen breath testing (H2BT) were published (meta-analysis by Varju 2019). This meta-analysis indicated that subjective LI was more frequently reported by IBS patients, but also objectively more prevalent in IBS patients, when assessed by any test modality. However, the role of a LFD in IBS remains uncertain.

This study aims to:

* Determine if the diagnosis of LM by H2BT predicts the short-term and long-term response to a LFD in moderate to severe IBS as defined by Rome IV criteria;
* Determine the changes in quality of life in response to a LFD in ROME IV IBS patients.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling the ROME IV criteria for IBS;
* Moderate symptom severity as defined by a IBS-SSS > 175;
* Consumption of lactose containing products.

Exclusion Criteria:

* Clinical suspicion of an organic disorder different from LI or IBS (patients can be included when this disorder had been excluded);
* Known lactose intolerance or malabsorption;
* Known inflammatory bowel disorder;
* Known intestinal motility disorder;
* Alcohol (defined as more than 14 U per week) or other substance abuse;
* Active psychiatric disorder;
* Known systemic or auto-immune disorder with implication for the GI system;
* Prior abdominal surgery (with the exception of appendectomy);
* Any prior diagnosis of cancer other than basocellular carcinoma;
* Current chemotherapy;
* History of gastro-enteritis in the past 8 weeks;
* Intake of antibiotics, pre- or probiotics during the past 8 weeks;
* Dietary supplements unless taken at a stable dose for more than 8 weeks;
* Treatment with neuromodulators (one neuromodulator taken at a stable dose for more than 12 weeks is allowed);
* Treatment with spasmolytic agents, opioids, loperamide, gelatin tannate or mucoprotect-ants during the past 8 weeks;
* LFD or low FODMAP diet in the past

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
symptomatic improvement | from baseline till visit 4 (week 4)
  To compare the symptomatic improvement by a LFD in Rome IV IBS patients with and without LM according to a H2BT.

SECONDARY OUTCOMES:
reduction in Irritable bowel syndrome - symptom severity scale | baseline till visit 4 (week 4)
  reduction in IBS-SSS at the end of 4 weeks of a LFD in Rome IV IBS subjects identified as lactose mal-absorbers vs. lactose absorbers by lactose H2BT

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No